CLINICAL TRIAL: NCT03808844
Title: A Multi-Center, Randomized, Double-Blind, Propofol-Controlled Phase III Clinical Trial Evaluating the Efficacy and Safety of HSK3486 Injectable Emulsion for the Induction of General Anesthesia in Elective Surgery Subjects
Brief Title: A Trial Evaluating the Efficacy and Safety of HSK3486 Injectable Emulsion for the Induction of General Anesthesia in Elective Surgery Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sichuan Haisco Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Organization: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSK3486-302
Record Dates: First submitted 2019-01-09; First posted 2019-01-18 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2018-12

CONDITIONS: Induction of Anesthesia
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HSK3486 (Experimental): 0.4mg/kg/0.2 mg/kg
  Interventions: Drug: HSK3486
- Propofol (Active Comparator): 2.0mg/kg/1.0mg/kg
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: HSK3486 — Initial dose of 0.4 mg/kg followed by 0.2 mg/kg if needed.
  Arms: HSK3486
Drug: Propofol — Initial dose of 2.0 mg/kg followed by 1.0 mg/kg if needed
  Arms: Propofol

SUMMARY:
This is a multi-center, randomized, double-blind, propofol-controlled phase III clinical trial. The primary objective is to compare the efficacy and safety between propofol and HSK3486 for the induction of general anesthesia in elective surgery subjects, so as to provide reference for marketing registration of HSK3486.

ELIGIBILITY:
Inclusion Criteria:

1. In-patients requiring tracheal intubation under general anesthesia for non-emergency, non-cardiothoracic, and non-extracerebral elective surgeries;
2. Male or female, ages between 18-64 (inclusive);
3. ASA (American Society of Anesthesiologists) Class I-II (see Appendix 4);
4. Body mass index (BMI) ≥18 and ≤30 kg/m2;
5. Vital signs: Respiratory rate ≥10 and ≤24 breaths per minute; blood oxygen saturation (SpO2) when inhaling ≥95%; systolic blood pressure (SBP) ≥90 mmHg and ≤160 mmHg; diastolic blood pressure (DBP) ≥60 mmHg and ≤100 mmHg; heart rate ≥55 and ≤100 bpm;
6. Subjects must understand the procedures and methods of this study, and be willing to provide informed consent and to complete the trial in strict accordance with study protocol.

Exclusion Criteria:

1. Patients with contraindications to general anesthesia or previous history of anesthesia accidents;
2. Known hypersensitivity to excipients and ingredients found in propofol and HSK3486 injections (soybean oil, glycerin, triglycerides, egg lecithin, sodium oleate, and sodium hydroxide), benzodiazepines, opioids, rocuronium bromide, sevoflurane, atropine, and neostigmine; cross-reactivity to halogenated anesthetics, jaundice or unexplained fever from previous use of halogenated anesthetics; contraindications to propofol;
3. Medical history or evidence of any of the following prior to screening/at baseline, which may increase sedation/anesthesia risk:

   1. History of cardiovascular diseases: Uncontrolled hypertension or SBP >160 mmHg and/or DBP >100 mmHg despite antihypertensive treatment, severe arrhythmia, heart failure, Adams-Stokes syndrome, unstable angina, myocardial infarction within 6 months before screening, history of tachycardia/bradycardia requiring medication, third-degree atrioventricular block or QTcF interval ≥450 ms (Fridericia's correction formula, see Appendix 2) during screening;
   2. Respiratory system disorders: Respiratory insufficiency, history of obstructive pulmonary disease, history of bronchospasm requiring treatment within 3 months prior to screening, acute respiratory tract infection with obvious symptoms such as fever, wheezing, or productive cough within 1 week prior to baseline;
   3. History of cerebrovascular disease: History of craniocerebral injury, convulsions, epilepsy, intracranial hypertension, cerebral aneurysm, or cerebrovascular accident; history of schizophrenia, mania, chronic use of antipsychotics, or cognitive impairment;
   4. Gastrointestinal disease history: Gastrointestinal retention, active hemorrhage, or circumstances that may lead to reflux and aspiration;
   5. Patient with a history of uncontrolled and clinically significant liver, kidney, blood system, nervous system or metabolic system diseases judged by the investigator to be unsuitable for this trial;
   6. History of alcohol abuse within 3 months prior to screening, abuse defined as average of >2 units of alcohol per day (1 unit = 360 mL beer or 45 mL liquor with 40% alcohol or 150 mL wine);
   7. History of drug abuse within 3 months prior to screening;
   8. Serious infection, trauma, or major surgery within 4 weeks prior to screening;
4. Any one of the following respiratory risks before/during screening:

   1. Asthma history, and stridor;
   2. Sleep apnea syndrome;
   3. History of malignant hyperthermia or family history;
   4. History of failed tracheal intubation;
   5. Judged by the investigator to have difficult airway or judged as difficult tracheal intubation (modified Mallampati score III or IV );
5. In receipt of any of the following drugs or therapies prior to screening:

   1. Participated in other drug trials within 1 month prior to screening;
   2. In receipt of medications that may affect QT interval within 2 weeks prior to screening (see Appendix 5);
   3. In receipt of medications that induce or inhibit cytochrome P450 isoenzyme CYP2B6 within 2 weeks prior to screening (see Appendix 6);
   4. In receipt of propofol, other sedatives/anesthetics, and/or opioid analgesics or compounds containing analgesics within 3 days prior to screening.
6. Laboratory results meeting any of the following criteria during screening/at baseline, confirmed by re-examination:

   1. Neutrophil count ≤1.5×109/L;
   2. Platelet count <80×109/L;
   3. Hemoglobin <90 g/L (no blood transfusion within the last 14 days);
   4. ALT and/or AST ≥2.0×upper limit of normal (ULN);
   5. Total bilirubin ≥2.0×ULN;
   6. Serum creatinine ≥1.5×ULN.
7. Women who are pregnant or breastfeeding; women of child-bearing potential or men who are unwilling to use contraception during the trial; subjects who are planning pregnancy within 1 month after the completion of the trial (including male subjects);
8. Subjects judged by the investigator to be unsuitable for participating in this trial for any reason.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 178 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
The success rate of induction of anesthesia | During induction of general anesthesia on day 1

SECONDARY OUTCOMES:
Time to successful anesthetic induction | From the initial administration of the investigational drug to the first time when MOAA/S is ≤1 on day 1
Time to loss of eyelash reflex | From the initial administration of the investigational drug to loss of eyelash reflex on day 1
Use of the investigational drug and alternative drugs | During induction of general anesthesia on day 1
Use of the alternative drugs | During induction of general anesthesia on day 1
Changes in bispectral index (BIS)（score：0~100） | During induction of general anesthesia on day 1
Number of patients with adverse events | Pre-dose to 48 hours post-dose
  Safety endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, China